CLINICAL TRIAL: NCT02684201
Title: Epidural Spinal Cord Stimulation for Sensory Restoration and Phantom Limb Pain in Upper-Limb Amputees
Acronym: PhantomLimb
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lee Fisher, PhD (Other)
Responsible Party: Sponsor-Investigator, Lee Fisher, PhD, PhD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19100220
Record Dates: First submitted 2015-11-11; First posted 2016-02-17 (Estimated); Results first posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Phantom Limb
Keywords: Phantom Limb; Upper Amputee; Electrodes; Implant; Pain
MeSH Terms: conditions — Phantom Limb; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Boston Scientific cord stimulator lead (Experimental): A Boston Scientific Stimulator Lead (PMA P030017) will be placed in the cervical epidural space of ten upper-limb amputees and steered laterally towards the dorsal spinal roots under fluoroscopic guidance.
  Interventions: Device: Boston Scientific Stimulator Lead

INTERVENTIONS:
Device: Boston Scientific Stimulator Lead — A Boston Scientific (PMA P030017) spinal cord stimulator lead will be placed in the cervical epidural space of ten upper-limb amputees and steered laterally towards the dorsal spinal roots under fluoroscopic guidance.

SUMMARY:
Individuals with upper-limb amputation usually have intact nerves within the residual limb, and studies have demonstrated that electrical stimulation of those nerves can produce sensations that appear to emanate from the amputated limb. In this study, investigators will examine the sensations that are produced by electrical stimulation of these nerves at the location where they exit the spinal cord. Stimulation of the spinal cord is commonly used to treat intractable back and limb pain, and the procedure includes a test phase in which electrodes are temporarily placed under the skin near the spinal cord and removed at the end of testing. Similarly, in this study, electrodes will be placed near the spinal cord in the upper back and neck, and stimulation will be applied over the course of multiple testing sessions, lasting less than 30 days. The electrodes will be removed at the last day of testing. During each testing session, electrical stimulation will be applied through the electrodes and a series of tests will be performed to determine the types of sensations produced by stimulation. In addition to producing meaningful sensations with electrical stimulation, this study will also test the effect of stimulation on phantom limb sensations and phantom limb pain.

DETAILED DESCRIPTION:
The purpose of this research study is to characterize the types of sensations that can be produced by stimulating the spinal nerves in upper-limb amputees, as well as the effects of that stimulation on phantom limb pain. The study involves a medical procedure to temporarily place one to three stimulation electrodes in the space near the spinal cord. This medical procedure will be performed under local anesthesia, and will take approximately one to two hours. Afterwards, the electrodes will be connected to an external stimulator and a series of experiments will be performed to characterize the types of sensations generated by electrical stimulation of the spinal cord and spinal nerves, as well as to measure the effect of stimulation on phantom limb sensations and phantom limb pain. Over the course of less than 30 days, there will be up to 20 of these experimental sessions. At the end of the final experimental session, the stimulation electrodes will be removed by gently pulling on them.

The investigators are inviting participants to consider participating in this research because they have an upper-limb amputation. Participants must be between the ages of 18 and 70 and at least one year post-amputation. Participants must be willing to travel to the University of Pittsburgh at least twice per week for 30 days.

Participants cannot have any serious diseases or disorders that affect your ability to participate in this study. Women who are pregnant or plan to become pregnant during the study cannot be included. The investigators will ask females of child-bearing potential to undergo a urine pregnancy test prior to any procedures (such as MRI, x-ray, fluoroscopy) that may disrupt the healthy development of an unborn child. If participants are currently taking any medications that thin their blood, participants will not be eligible for this study. Participants will have to meet other criteria to be eligible, which will be reviewed with participants upon their consent. The investigators will screen up to 15 people and expect that up to 10 individuals will complete this study.

ELIGIBILITY:
Inclusion Criteria:

* have an upper-limb amputation
* must be between the ages of 18 and 70
* be at least one year post-amputation
* be willing to travel to the University of Pittsburgh at least twice per week for 29 days

Exclusion Criteria:

* women who are pregnant or plan to become pregnant during the study
* all participants cannot have any serious diseases or disorders that affect your ability to participate in this study
* must not be currently taking any medications that thin your blood

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee E Fisher, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Study sponsors will have access to research data and documents in order to monitor the integrity of the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Study information will be shared with the study sponsor through the duration of the grant.
Access Criteria: Data will be shared with the sponsor and/or collaborators per the stipulations of the grant and/or data sharing agreements.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were met in amputee clinics, referred by prosthetics representatives, or responded to advertisements posted at amputee support groups. The study team spoke with approximately 25 interested patients. Of these, four completed the consent process.
Pre-assignment Details: Eligibility checking ruled out participants due to congenital missing limb (not amputation), taking prescription blood thinners, or unable to refrain from physical exertion during the duration of the experiment. These individuals were either excluded, or withdrew. Others declined the surgery.
Period: Overall Study
Arm/Group | Boston Scientific Cord Stimulator Lead
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The first participant experienced lead migration and early explant. This participant was later re-enrolled and completed study activities. Therefore, there are 4 unique individuals counted among the 5 consented participants.
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4
Participants with phantom limb pain [Count of Participants; unit: Participants] — Participants who report having phantom limb pain
  Participants | 3

OUTCOME MEASURES:

1. Primary Outcome: Stimulation Thresholds to a Variety of Stimulus Parameters
Description: Quantify the threshold (minimum charge) stimulus required to evoke sensation and neurophysiological responses during epidural spinal nerve stimulation, and monitor changes in those percepts and responses over time.
Time Frame: 30 days
Population: Participants implanted with stimulator leads
Measure: Mean (Full Range); unit: milliamps
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 4
milliamps | 2.13 [1.25 to 3.75]

2. Primary Outcome: Week 1 Average Stimulus Charge for All Subjects
Description: The average stimulus (nC) required to evoke sensation during week 1 of implant duration.
Time Frame: first 7 days of implant
Measure: Mean (Full Range); unit: nC
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 4
nC | 647 [174 to 4000]

3. Primary Outcome: Week 2 Average Stimulus Charge for All Subjects
Description: The average stimulus (nC) required to evoke sensation during week 2 of implant duration.
Time Frame: During days 7-14 of implant
Measure: Mean (Full Range); unit: nC
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 4
nC | 807 [300 to 4384]

4. Primary Outcome: Week 3 Average Stimulus Charge for All Subjects
Description: The average stimulus (nC) required to evoke sensation during week 3 of implant duration.
Time Frame: During days 15 to 21 of implant
Population: Participant 2 had the stimulator removed before week 3. Participants 1, 3, and 4 were included in this analysis.
Measure: Mean (Full Range); unit: nC
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 3
nC | 1115 [500 to 4800]

5. Primary Outcome: Week 4 Average Stimulus Charge for All Subjects
Description: The average stimulus (nC) required to evoke sensation during week 4 of implant duration.
Time Frame: During days 22-28 of implant
Population: Participant 2 had the stimulator removed before week 3. Participants 1, 3, and 4 were included in this analysis.
Measure: Mean (Full Range); unit: nC
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 3
nC | 902 [300 to 3775]

6. Secondary Outcome: Number of Participants Who Were Able to Discern Specific Regions of the Spinal Cord That Evoked Sensations
Description: Evaluate the relationship between stimulation parameters and the modality and naturalness of perceived sensations.
Time Frame: 30 days
Population: Participants with implanted spinal cord stimulator who were able to discern specific regions of the spinal cord that evoked sensations
Measure: Count of Participants; unit: Participants
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 4
Participants
  Felt stimulation | 4
  Felt stim in hand | 4
  Felt stim in elbow | 3
  Felt stim in shoulder | 2
  Felt stim in fingers | 4
  C6 evoked stim | 3
  C7 evoked stim | 3
  C8 evoked stim | 4
  T1 evoked stim | 4
  T2 evoked stim | 2

7. Secondary Outcome: Qualitative Self-report of Evoked Sensations
Description: Document the subjective perception of cervical epidural spinal nerve stimulation for restoration of sensation. The investigators will ask each subject to provide subjective feedback on their perceived utility of the sensory feedback provided by the device.
Time Frame: 30 days
Population: Participants implanted with spinal cord stimulator who reported sensations felt
Measure: Count of Participants; unit: Participants
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 4
Participants
  Paresthetic sensation (primarily) | 1
  Mixed Modality (paresthetic and naturalistic) | 2
  Naturalistic (primarily) | 1

8. Secondary Outcome: Change in Pain Ratings After Study Completion
Description: Participants were asked to complete the McGill pain questionnaire at baseline, and weekly throughout implant. We expected to see a decrease in the pain level due to electrical stimulation. A positive score indicates a decrease in level of pain (baseline - study end). Minimum score is 0. Maximum score is 80. The higher the number, the greater the pain. This outcome measure suntracts the baseline pain score from the final pain score. A positive score indicates a reduction in pain from baseline.
Time Frame: 30 days
Population: Participants were asked to complete the McGill pain questionnaire at baseline, and weekly throughout implant. We expected to see a decrease in the pain level due to electrical stimulation. A positive score indicates a decrease in level of pain (baseline - study end). Three participants reported having phantom limb pain prior to the study.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Boston Scientific Cord Stimulator Lead
Number analyzed (Participants) | 3
score on a scale
  Change in Pain Score (baseline - final) | 14.3 [6 to 20]
  Baseline Pain Score | 32.3 [29 to 35]
  Final Pain Score | 18 [12 to 29]

9. Secondary Outcome: Success Rate During Control of Prosthetic Hand to Identify Object Size
Description: Investigators will test the subject's ability to use a myoelectric prosthetic hand with and without sensory feedback provided by electrical stimulation of the spinal roots. Using either a virtual prosthetic limb or an instrumented prosthesis, stimulation of the spinal roots will be modulated based on signals recorded from the limb such as pressure at the finger tips or joint angles. In both the presence and absence of stimulation, subjects will be asked to perform tasks such as manipulating blocks, opening a jar, or identifying the stiffness and size of various objects.
Time Frame: 30 days
Population: Person with upper limb amputation for over two years. This subject had a high trans-humeral amputation and did not have sufficient musculature in the residual limb to achieve reliable myoelectric control of the prosthesis. Instead, she wore a Data Glove (Fifth Dimension Technologies, 5 DT) on her contralateral, intact hand, and the grasp aperature from the Data Glove was used to proportionally control the aperture of the real and cirtual DEKA hand.
Measure: Number; unit: percentage of success identifying size
Groups:
- Size Discrimination Using Virtual DEKA Arm: Presented with four different sizes of cubes: extra small, small, medium, and large, all from the same foam rubber material. Presentation order was randomized and subject did not have visual feedback. Subject did not explore an object for more than 10 seconds.
Arm/Group | Size Discrimination Using Virtual DEKA Arm
Number analyzed (Participants) | 1
percentage of success identifying size | 74

10. Secondary Outcome: Success Rate During Control of Prosthetic Hand to Identify Object Compliance (Soft, Medium, Hard)
Description: Investigators tested the subject's ability to use a myoelectric prosthetic hand with and without sensory feedback provided by electrical stimulation of the spinal roots. Using either a virtual prosthetic limb or an instrumented prosthesis, stimulation of the spinal roots was modulated based on signals recorded from the limb such as pressure at the finger tips or joint angles. In both the presence and absence of stimulation, subjects were asked to perform tasks such as manipulating blocks, opening a jar, or identifying the stiffness (soft, medium, hard) and size of various objects.
Time Frame: 30 days
Population: Person with upper limb amputation for over two years. This subject had difficulty achieving reliable prosthesis control, even with simple control schemes such as parallel dual-site control. As such, a highly simplified control scheme was implemented, in which the subject was instructed to attempt a hand grasp, and when this signal crossed a manually defined threshold, the DEKA hand was commanded to close at a constant velocity of 15 degrees/second.
Measure: Number; unit: percentage of success identifying compli
Groups:
- Compliance Discrimination Using DEKA Arm: Presented with cylinders of three different sizes (small, medium, and large), and three different compliances (soft, medium, and hard). Presentation order was randomized and subject did not have visual feedback or audio.
Arm/Group | Compliance Discrimination Using DEKA Arm
Number analyzed (Participants) | 1
percentage of success identifying compli | 60

ADVERSE EVENTS:
Time Frame: 30 days (duration of implant)
Arm/Group | Boston Scientific Cord Stimulator Lead
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Boston Scientific Cord Stimulator Lead (N=4)
Lead migration (Surgical and medical procedures) | 2 — Movement of spinal cord lead(s) after implant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-01-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT02684201/Prot_SAP_000.pdf